CLINICAL TRIAL: NCT06868810
Title: Comparison of 5% Sodium Bicarbonate and 10% Sodium Chloride As Contrast Agents for Lung Perfusion with Electrical Impedance Tomography: a Prospective Clinical Study
Brief Title: Comparison of 5% Nacl and 10% NaHCO3 As Contrast Agents for Lung Perfusion with EIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EIT contrast agent
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
MeSH Terms: conditions — Acute Lung Injury | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NaCl (Experimental): First, perform the EIT contrast method with 10% NaCl. After a 10-minute washout period, perform the EIT contrast method with 5% NaHCO3.
  Interventions: Other: Injection of hypertonic saline; Other: Injection of 5% NaHCO3
- NaHCO3 (Other): First, perform the EIT contrast method with 5% NaHCO3. After a 10-minute washout period, perform the EIT contrast method with 10% NaCl.
  Interventions: Other: Injection of hypertonic saline; Other: Injection of 5% NaHCO3

INTERVENTIONS:
Other: Injection of hypertonic saline — Injection 10 mL of 10% NaCl through central venous catheter
Other: Injection of 5% NaHCO3 — Injection of 5% NaHCO3 through central venous catheter

SUMMARY:
Electrical impedance tomography (EIT) has enabled the bedside monitoring of lung perfusion measurement through the indicator-based contrast method. Currently, hypertonic sodium chloride is the most commonly used contrast agent for lung perfusion evaluation by EIT. However, concerns may be raised regarding the potential risks of hyperchloremia and possible acute kidney injury associated with the use of hypertonic NaCl. Recently, two experimental studies found sodium bicarbonate (NaHCO3) might be an alternative to hypertonic sodium chloride in lung perfusion assessment by EIT. However, whether NaHCO3 results in acceptable bias is unknown in critically ill patients. This clinical study aimed to further investigate the correlation and agreement of lung perfusion and Ventilation/perfusion (V/Q) match by EIT contrast method between two contrast indicators (5%NaHCO3 vs. 10% NaCl) in critically ill patients with respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* In need of lung perfusion assessment due to clinical condition
* With central venous catheter

Exclusion Criteria:

* contraindications to the use of EIT (automatic implantable cardioverter defibrillator, chest wounds limiting electrode belt placement, implantable pumps, etc.)
* severe hyperchloremia (>155 mmol/L)
* unable to tolerate breath-hold maneuver
* pregnant or breastfeeding females

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
lung perfusion distribution in ROI | Offline analysis, immediately after the saline injection procedure

SECONDARY OUTCOMES:
V/Q match in ROI | Offline analysis, immediately after the saline injection procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided